CLINICAL TRIAL: NCT02836366
Title: Prospective Cohort Study of Proximal Humeral Fractures Treated With Targon® PH+
Brief Title: Targon PH+ Follow-Up
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1536
Record Dates: First submitted 2016-06-10; First posted 2016-07-19 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Shoulder Fractures
Keywords: Proximal humerus; Fracture; Nailing
MeSH Terms: conditions — Shoulder Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
With this study results of the Targon® PH+ nail, developed for the treatment of humeral head fractures, will be investigated clinically, radiological evaluation is optional. The primary objective of this study is to examine the effect of a plating treatment on the speed of recovery of functional capacity in adult patients. Secondary aims are to examine the level of pain, patient satisfaction, shoulder function, quality of life, radiological evaluation and complications.

Targon PH+ is CE certified. The study is a non-interventional cohort study sponsored by Aesculap

ELIGIBILITY:
Inclusion Criteria: - patients with a three- or four-fragment-fracture of the proximal humerus, with dislocation on X-ray

* older than 60 years of age
* written and signed patient consent

Exclusion Criteria: - Fractures more than 14 days old

* multiple comorbidity
* multitrauma (Injury Severity Score > 15)
* prev. surgery on the injured shoulder
* severely deranged function caused by a previous disease head-split proximal humerus fracture
* combined humerus head and shaft fractures
* pseudarthroses
* crushed head cap of the humerus head (AO 11 C3 fractures)
* isolated avulsion fracture of a tuberosity
* unwillingness or inability to follow protocol instructions and study requirements (follow-up visits)
* no signed informed consent
* treatment not in line with Instructions for Use (IfU)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Functional Capacity | 24 months
  The DASH score (Disabilities of the Arm, Shoulder, and Hand) will be used to determine the recovery of functional capacity. It provides a summary of the responses on a scale of 0 (no disability) to 100 (severe disability)

SECONDARY OUTCOMES:
Level of pain | 3, 12 and 24 months
  10-point Visual Analogue Scale (VAS) from no pain (0) to most extreme pain imaginable (10)
Patient satisfaction | 24 months
  4 point scale: very satisfied, satisfied, unsatisfied, very unsatisfied
Shoulder Function | 12 months, 24 months
  Shoulder function outcome is measured with the Constant-Murley score, this score system combines shoulder function tests (65 points) with a subjective evaluation of the patients (35 points) including activities of daily living, level of work
Radiological outcome (only if it could be raised in clinical standard) | 24 months
  The X-rays are examined regarding adverse events as screw perforation, screw breakage, cut-out, re-dislocation of the fracture
Adverse Events | 24 months
  Rate of Adverse Events, for example secondary interventions (revisions) that occur within the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Hermann Josef Bail, Prof. Dr., Principal Investigator — Klinikum Nürnberg Süd
Locations (1):
- Klinikum Nürnberg Süd, Nuremberg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No